CLINICAL TRIAL: NCT03743961
Title: Description the Geriatric Intervention Contribution on Quality of Life of Elderly Patients With Metastatic Neoplasia : Prospective Descriptive Non-comparative Cohort ( QUALI Cohort)
Brief Title: Geriatric Intervention Contribution on Quality of Life of Elderly Patients With Metastatic Neoplasia
Acronym: QUALI
Status: Terminated | Type: Observational
Why Stopped: Low rythm of inclusions
Sponsor: Institut de Cancérologie de la Loire (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-0801; 2018-A02315-50 (Other: ANSM)
Record Dates: First submitted 2018-10-08; First posted 2018-11-16 (Actual); Last update posted 2020-07-07 (Actual); Status verified 2020-07

CONDITIONS: Systemic Treatment; Metastatic Neoplasia; Elderly Patients
Keywords: quality of life; elderly; metastatic neoplasia; systemic therapies
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group A : control group: Evaluation of quality of life with the EORTC QoL ELD 14 (Quality Qf Life ELDerly patients with 14 Questions) and QoL EORTC Q30 (Quality Qf Life with 30 Questions)
  for patients with G8 score > 14/17
- Group B : geriatric intervention group: Evaluation of quality of life with the EORTC QoL ELD 14 (Quality Qf Life ELDerly patients) and QoL (Quality Qf Life) EORTC Q30 for patients with G8 score ≤14/17 ( in this arm there is two groups : patient who received geriatric intervention before treatment initiation (group A) and group of patient did not received geriatric intervention before treatment initiation( group B))
  Interventions: Other: geriatric intervention

INTERVENTIONS:
Other: geriatric intervention — Geriatric intervention
  Groups: Group B : geriatric intervention group

SUMMARY:
The aim of this study is to describe the impact of : Geriatric intervention contribution on quality of life of elderly patients receiving systemic treatments for metastatic neoplasia

DETAILED DESCRIPTION:
Elderly cancer incidence increases exponentially with advancing age. However, elderly patients are largely underrepresented in cancer treatment trials. The geriatric population presents particular physical, mental, psychological or social specificities that may condition the prognosis especially for patients with metastatic neoplasia. Recently, the measurement of quality of life (QoL) in aging population is being recognized as an important part of clinical decision. It is therefore essential to set up prospective studies to evaluate the impact of oncogeriatric practices on the quality of life of elderly patients with metastatic neoplasia. The main objective of this prospective study is to describe the contribution of geriatric intervention on quality of life for for elderly (> 75 years) with metastatic solid cancer receiving systemic treatment during the first 6 months of their therapeutic management.

ELIGIBILITY:
Inclusion Criteria:

* Patient with solid metastatic neoplasia
* 75 years old or more
* Men or women
* ECOG between 0 and 3
* Patient receiving systemic antineoplasic treatment (chemotherapy, hormonotherapy, immunotherapy, targeted therapy)

Exclusion Criteria:

* ECOG 4
* Localized cancer
* Patients already included in a study witch could modify quality of life
* Patient unable to give their consent

Min Age: 75 Years | Sex: All
Age Groups: Older Adult
Study Population: Patients with minimum 75 years old will perform two questionnaires about quality of life and then, according to these scores they will perform a geriatric intervention.
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-11-21 (Actual); Primary Completion 2020-07-02 (Actual); Study Completion 2020-07-02 (Actual)

PRIMARY OUTCOMES:
Level of quality of life | 6 months
  Level of quality of life will be measured with the QoL ELD 14 (Quality Qf Life ELDerly patients with 14 Questions)
Level of quality of life | 6 months
  Level of quality of life will be measured with the QoL Q30 (Quality Qf Life with 30 Questions)

SECONDARY OUTCOMES:
number of hospitalizations | 6 months
  number of hospitalizations will be reported
Duration of hospitalizations | 6 months
  Duration of hospitalizations will be reported in hours
Number of toxicities ( grade 3 and 4) | 6 months
  Number of toxicities (grade 3 and 4) will be reported according to the CTCAE v4.0 (Common Terminology Criteria for Adverse Events)

CONTACTS AND LOCATIONS:
Overall Officials: Blandine De Lavigerie, MD, Principal Investigator — Institut de Cancérologie Lucien Neuwirth
Locations (1):
- Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez, France

IPD SHARING:
Plan to Share IPD: No